CLINICAL TRIAL: NCT01008189
Title: 6-Year Follow-up of a Prevention Program for Bereaved Families
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Irwin Sandler, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH049155 (NIH); R01MH049155 (NIH)
Record Dates: First submitted 2009-09-24; First posted 2009-11-04 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Mental Disorders Diagnosed in Childhood
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self study comparison group (Active Comparator): Caregivers and children and adolescents each received three books about coping with grief after the death of a loved one and a syllabus to guide reading
  Interventions: Behavioral: Self- study comparison group
- Family Bereavement Program (Experimental): 12- session group for caregivers and bereaved children and adolescents plus 2 individual sessions
  Interventions: Behavioral: Family Bereavement Program

INTERVENTIONS:
Behavioral: Self- study comparison group — Caregivers, children and adolescents each received three books about coping with grief following the death of a loved one plus a syllabus to guide reading
  Arms: Self study comparison group
Behavioral: Family Bereavement Program — 12 session groups for caregivers and bereaved children and adolescents plus two individual sessions
  Arms: Family Bereavement Program

SUMMARY:
Six-years following participation in the Family Bereavement Program (FBP) participants in the program as compared to a self-study control group will have lower levels of mental health problems, lower one-year prevalence of mental disorder that meets diagnostic criteria, lower use of substances, higher levels of competence at achieving developmentally appropriate tasks in academic achievement and social competence, and better self-esteem. The effects of the FBP will be moderated by baseline levels of mental health problems and gender. Bereaved caregivers who participated in the program will also show lower levels of mental health problems as compared with controls.

Program effects will be mediated by theoretical mediators targeted by the program.

ELIGIBILITY:
Inclusion Criteria:

* Experienced parental death in prior 30 months
* Youth age 8-16 years old

Exclusion Criteria:

* Not currently in other treatment for mental health problems
* Caregiver not meet criteria for clinical depression
* Youth not meet criteria for externalizing problems
* Not currently suicidal

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 1996-01; Primary Completion 2005-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic Interview Schedule for Children (DISC) | One year
Child Behavior Checklist and Young Adult Behavior Checklist | one year
Youth Self Report (YSR)and Young Adult Self Report (YASR) | one year

SECONDARY OUTCOMES:
Monitoring the Future - substance use | one year
Rosenberg Self-esteem scale | one year
Beck Depression Inventory for parents | One week
Social and academic competence | one year
Grade point average | one year
Cortisol | 45 minutes
Parent and child report of parenting | One year
Grief - TRIG, Intrusive Grief Thoughts Scale, Inventory of Complicated Grief | one month

CONTACTS AND LOCATIONS:
Overall Officials: Irwin N Sandler, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Prevention Research Center Arizona State University, Tempe, Arizona, United States

REFERENCES:
- [Background] Sandler IN, Ayers TS, Wolchik SA, Tein JY, Kwok OM, Haine RA, Twohey-Jacobs J, Suter J, Lin K, Padgett-Jones S, Weyer JL, Cole E, Kriege G, Griffin WA. The family bereavement program: efficacy evaluation of a theory-based prevention program for parentally bereaved children and adolescents. J Consult Clin Psychol. 2003 Jun;71(3):587-600. doi: 10.1037/0022-006x.71.3.587. PMID 12795581
- [Derived] Sandler I, Tein JY, Zhang N, Wolchik SA. Developmental Pathways of the Family Bereavement Program to Prevent Major Depression 15 Years Later. J Am Acad Child Adolesc Psychiatry. 2023 Nov;62(11):1233-1244. doi: 10.1016/j.jaac.2023.02.012. Epub 2023 Mar 8. PMID 36898606
- [Derived] Danvers AF, Scott BG, Shiota MN, Tein JY, Wolchik SA, Sandler II. Effects of Therapeutic Intervention on Parentally Bereaved Children's Emotion Reactivity and Regulation 15 Years Later. Prev Sci. 2020 Nov;21(8):1017-1027. doi: 10.1007/s11121-020-01142-2. PMID 32720190
- [Derived] Sandler I, Tein JY, Cham H, Wolchik S, Ayers T. Long-term effects of the Family Bereavement Program on spousally bereaved parents: Grief, mental health problems, alcohol problems, and coping efficacy. Dev Psychopathol. 2016 Aug;28(3):801-18. doi: 10.1017/S0954579416000328. PMID 27427807
- [Derived] Sandler I, Ayers TS, Tein JY, Wolchik S, Millsap R, Khoo ST, Kaplan D, Ma Y, Luecken L, Schoenfelder E, Coxe S. Six-year follow-up of a preventive intervention for parentally bereaved youths: a randomized controlled trial. Arch Pediatr Adolesc Med. 2010 Oct;164(10):907-14. doi: 10.1001/archpediatrics.2010.173. PMID 20921347